CLINICAL TRIAL: NCT04714268
Title: Comparison of Aorto-iliac Endovascular Interventions With and Without the EndoNaut Workstation
Acronym: COM-ENDO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Therenva (Industry)
Collaborators: Rennes University Hospital (Other); Douai hospital (Unknown); Centre Hospitalier Universitaire Dijon (Other); University Hospital, Brest (Other); Polyclinique Bordeaux Nord Aquitaine (Other)
Responsible Party: Sponsor
Other Study IDs: 002
Record Dates: First submitted 2021-01-15; First posted 2021-01-19 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Aortic Aneurysm; Iliac Aneurysm; Stenoses, Aortic; Iliac Artery Stenosis
MeSH Terms: conditions — Aortic Aneurysm; Iliac Aneurysm; Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Procedures with EndoNaut: Endovascular interventions using the EndoNaut workstation. 3D image fusion is used for overlaying arterial information on top of fluoroscopic images
  Interventions: Procedure: Aorto-iliac endovascular procedure
- Procedures without EndoNaut: Control group, endovascular interventions without 3D image fusion
  Interventions: Procedure: Aorto-iliac endovascular procedure

INTERVENTIONS:
Procedure: Aorto-iliac endovascular procedure — Percutaneous procedure with stent placement

SUMMARY:
The aim of this retrospective, multicenter study is to demonstrate that the use of EndoNaut for aortoiliac endovascular procedures has a clinical impact for the patient (reduction in irradiation and the volume of contrast product) as well as for the nursing staff (reduction irradiation) compared to procedures performed without EndoNaut.

DETAILED DESCRIPTION:
Minimally invasive endovascular interventions are increasingly replacing conventional surgeries, and have become the therapeutic benchmark for a large number of pathologies thanks in particular to advances in image-guided therapy. Therenva offers a comprehensive and consistent lightweight navigation solution (EndoNaut®) for endovascular procedures. This navigation station makes it possible to secure and guide the interventional gesture by providing relevant information extracted during the preoperative phase. This information is rendered in augmented reality using artificial intelligence algorithms and digital simulation. This alternative solution to a hybrid room, but which offers equivalent functionality, is compatible with all operating rooms, regardless of the interventional environment. Benefits of imaging fusion remain to be assessed on a larger scale. The aim of this multicenter study is to demonstrate that the use of EndoNaut for aortoiliac endovascular procedures has a clinical impact for the patient (reduction in irradiation and the volume of contrast product) as well as for the nursing staff (reduction irradiation) compared to procedures performed without EndoNaut.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral or bilateral aorto-iliac or iliac aneurysm/stenosis
* Suitable for endovascular repair
* Major patients
* Patients not opposed to their participation in the study

Exclusion Criteria:

* Patients requiring conventional surgical revascularization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female patients with unilateral or bilateral common iliac aneurysm or stenosis, treated with endovascular technique
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Volume of contrast product used during the routine care procedure (ml) | At enrollment
  Volume are reported in mL
Irradiation parameters: evaluation of the Fluoroscopy duration (min) | At enrollment
  Parameter given by the X-ray imaging device
Irradiation parameters: dose-area quantification (mGy/m2) | At enrollment
  Parameter given by the X-ray imaging device
Irradiation parameters: measurement of air Kerma (mGy) | At enrollment
  Parameter given by the X-ray imaging device

SECONDARY OUTCOMES:
Procedure time (min) | At enrollment
  Total procedure time

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Rennes, Rennes, France

IPD SHARING:
Plan to Share IPD: No